CLINICAL TRIAL: NCT03963466
Title: A Randomized Controlled Trial of the Efficacy and Safety of 1064-nm Q-Switched Fractional Laser Combined With Oral Tranexamic Acid on Treating of Melasma.
Brief Title: A Clinical Observation of 1064-nm Q-Switched Fractional Laser Combined With Oral Tranexamic Acid on Treating of Melasma.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: xjpfW (Other)
Collaborators: Air Force General Hospital of the PLA (Other Government); First Hospital of China Medical University (Other); Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, xjpfW, Head of Dermatology, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: XijingH-PF-20190430
Record Dates: First submitted 2019-05-10; First posted 2019-05-24 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Melasma
Keywords: Melasma; 1064-nm Q-Switched Fractional Laser; Tranexamic acid (TA); Treatment
MeSH Terms: conditions — Melanosis | interventions — Tranexamic Acid; Lasers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group 1 (Experimental): (left side of cheek) 1064-nm Q-Switched fractional laser+drug Device: 1064-nm Q-Switched fractional laser is used for melisma with the MASI ≥24 Drug: Oral tranexamic acid group(menstrual period>2days)
  Interventions: Drug: tranexamic acid; Radiation: 1064-nm Q-Switched fractional laser
- group 2 (Experimental): (right side of cheek) 1064-nm Q-Switched laser+drug Device: 1064-nm Q-Switched laser is used for melisma with the MASI ≥24 Drug: Oral tranexamic acid group(menstrual period>2days)
  Interventions: Drug: tranexamic acid; Radiation: 1064-nm Q-Switched laser
- group 3 (Experimental): (left side of cheek) 1064-nm Q-Switched fractional laser Device: 1064-nm Q-Switched fractional laser is used for melisma with the MASI ≥24
  Interventions: Radiation: 1064-nm Q-Switched fractional laser
- group 4 (Experimental): (right side of cheek) 1064-nm Q-Switched laser Device: 1064-nm Q-Switched laser is used for melisma with the MASI ≥24
  Interventions: Radiation: 1064-nm Q-Switched laser

INTERVENTIONS:
Drug: tranexamic acid — Oral tranexamic acid group(menstrual period>2days) 250mg bid（exclude menstrual period ）
  Arms: group 1; group 2
Radiation: 1064-nm Q-Switched fractional laser — Device: 1064-nm Q-Switched fractional laser is used for melisma with the MASI ≥24 left side of cheek is selected to be treated with 1064-nm Q-Switched fractional laser therapy (8ms, 1.5±0.5J/cm2) once 4 weeks for a total of 5 times
  Arms: group 1; group 3
Radiation: 1064-nm Q-Switched laser — Device: 1064-nm Q-Switched laser is used for melisma with the MASI ≥24 right side of cheek is selected to be treated with 1064-nm Q-Switched laser therapy (8ms, 1.5±0.5J/cm2) once 4 weeks for a total of 5 times
  Arms: group 2; group 4

SUMMARY:
1.Melasma is a common acquired condition of symmetric hyperpigmentation, typically occurring on the face, with higher prevalence in females and darker skin types. Treatments for melasma include topical, oral, procedural, and combination treatments.

2.1064-nm Q-Switched laser is one of the most widely used lasers for pigmented diseases in recent years. This wavelength laser can be effectively absorbed by pigment, which leads to damage of pigment and melanocyte. Previous 1064-nm Q-Switched laser treatment of melasma requires the use of large flare and low energy scanning repeatedly in the lesion area, and the terminal reaction is reddish and skin lesion temperature increased by 2℃. So the course of treatment is even longer and is closely related to the treatment of the doctor's subjective judgment. Current 1064-nm Q-Switched fractional laser is designed with focusing lens and can be scanned only once for skin lesions during treatment. Further more, the treatment energy of a single point is higher and it has stronger ability to destroy melanin. Finally, 1064-nm Q-Switched fractional laser promotes the expulsion of melanin particles from the superficial dermis and basal epidermis.

3.Tranexamic acid (TA) works by inhibiting the plasmin-plasminogen pathway. Increase in plasmin in keratinocytes leads to increase in production of arachidonic acid and alpha-melanocyte-stimulating hormone (alpha-MSH) production. Thus, by inhibiting the plasmin pathway, TA results in decreased melanogenesis. Studies support the use of oral TA as an adjuvant therapy for in refractory cases of melasma or as a second-line or third-line agent, and there is some early evidence supporting the utility of oral TA as monotherapy. Overall, randomized controlled trials have found that combination treatment regimens using oral TA as adjunct therapy results in greater reduction of melasma.

ELIGIBILITY:
Inclusion Criteria:

.Subjects must be clinically diagnosed by the investigator to melasma and MASI score ≥24.

* no other treatment was performed for the skin lesions for half a year before the treatment
* (patients with a "no" in any of the above criteria are not eligible for inclusion) .Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures being conducted.

Exclusion Criteria:

* subjects with a recent history of exposure to sunlight;
* subjects allergic to topical anesthesia;
* subjects with scar constitution;
* subjects with skin malignant tumors or precancerous lesions; .subjects with diabetes, heart disease, epilepsy, connective tissue disease, etc.
* subjects who Pregnant or breast feeding;
* subjects with recent skin infections (such as viruses, bacteria, etc.);
* the methods are being used to treat subjects with similar diseases;
* subject who have taken isotretinoin A in the past year; .subject with facial dermatitis.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Melasma area and severity index (MASI) | From 0weeks to 36Weeks
  Quantitative analysis was made according to the area, depth and uniformity of melasma. Pigmentation area was assessed in four areas: the forehead (F) 30%, the right cheek (MR) 30%, the left cheek (ML) 30%, and the mandible (C) 10%. According to the proportion of pigmented spots in the four areas, the scores were: 1 was less than 10%, 2 was 10%-29%, 3 was 30%-49%, 4 was 50%-69%, 5 was 70%-89%, 6 was 90%-100%. Color Depth (D) and Uniformity (H) Scores: 0 - 4 points: 0 points for none, 1 points for slight, 2 points for moderate, 3 points for obvious, 4 points for maximum. MASI = forehead [0.3A (D + H)] + right cheek [0.3A (D + H)] + left cheek [0.3A (D + H)] + mandible [0.1A (D + H)]. The maximum score is 48 and the minimum is 0.
Antera 3D skin test | From 0weeks to 36Weeks
  Antera 3D skin test measures the changes of skin melanin and hemoglobin before and after treatment quantitatively.
VISIA image analysis system | From 0weeks to 36Weeks
  VISIA image analysis system: different light sources, such as standard, ultraviolet and orthogonal polarization, are used to quantify different skin states. The patients with melasma are judged the number, distribution, area, depth and capillary condition of pigments by surface, ultraviolet and brown spots.

SECONDARY OUTCOMES:
Patient self-evaluation | 20Weeks，36Weeks
  Through questionnaires, patients' satisfaction with curative effect was investigated, which was divided into very satisfactory (improvement (> 75%), satisfactory (improvement 50% - 75%), general (improvement 25% - 50%) and unsatisfactory (improvement (< 25%). Statistical satisfaction rate was obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, Prof, Principal Investigator — Dermatology Derpartment of Xijing Hospital
Locations (1):
- Dermatology Derpartment of Xijing Hospital, Xi'an, Shaanxi, China